CLINICAL TRIAL: NCT01398943
Title: Regulation of Nitric Oxide Bioavailability in Chronic Obstructive Pulmonary Disease: A Mechanistic Approach
Brief Title: Nitric Oxide Bioavailability in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ryan Harris, Assistant Professor, Director Laboratory of Integrative Vascular and Exercise Physiology, Augusta University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AHA00115CS
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: flow-mediated dilation; arterial stiffness; intima-media thickness; pulse wave velocity; dual energy x-ray absorptiometry; inflammatory markers; blood lipids; tetrahydrobiopterin; body mass index; hemoglobin A1c; complete blood count; oxidative stress biomarkers; pulmonary function test; lung; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD Patients (Experimental): Patients with COPD
  AOC protocol: Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) will be assessed at baseline and 2 hours following ingestion of a single oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid
  BH4 protocol: Brachial artery flow-mediated dilation (FMD), markers of inflammation, and markers of oxidative stress will be assessed at baseline and following an increase in nitric oxide bioavailability after administering a single dose = 5 mg/kg of Tetrahydrobiopterin (BH4)
  Interventions: Drug: Tetrahydrobiopterin (BH4); Dietary Supplement: Antioxidant Cocktail
- Controls (Experimental): Healthy age- and sex- matched controls
  AOC protocol: Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) will be assessed at baseline and 2 hours following ingestion of a single oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid
  BH4 protocol: Brachial artery flow-mediated dilation (FMD), markers of inflammation, and markers of oxidative stress will be assessed at baseline and following an increase in nitric oxide bioavailability after administering a single dose = 5 mg/kg of Tetrahydrobiopterin (BH4)
  Interventions: Drug: Tetrahydrobiopterin (BH4); Dietary Supplement: Antioxidant Cocktail

INTERVENTIONS:
Drug: Tetrahydrobiopterin (BH4) — single dose = 5 mg/kg
  Other Names: Kuvan (Sapropterin Dihydrochloride)
Dietary Supplement: Antioxidant Cocktail — 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid

SUMMARY:
More patients with chronic obstructive pulmonary disease (COPD) die from cardiovascular disease than direct pulmonary complications. Inflammation and oxidative stress, characteristic in COPD, are likely contributors to the reduction in nitric oxide (NO) bioavailability and vascular endothelial dysfunction in COPD patients; however, this has yet to be determined. Thus, the overall objective of this proposal is to identify the role of NO bioavailability in contributing to vascular endothelial dysfunction in patients with COPD and to provide insight into the molecular mechanisms involved. Our central hypothesis is that inflammation and oxidative stress, both independently, contribute to the reduction in NO bioavailability and vascular endothelial dysfunction in patients with COPD.

DETAILED DESCRIPTION:
Flow-Mediated Dilation (FMD) - Subjects will lie in the supine position for 20 minutes to obtain hemodynamic steady state. A blood pressure cuff (Hokanson) will be placed around the forearm (distal to the Doppler transducer) and rapidly inflated to 250 mmHg for 5 minutes (circulatory arrest). Simultaneous ultrasound images of the vessel (B-mode) and Doppler waveforms will be collected 10 seconds prior to and for 2 minutes following deflation of the cuff. All B-mode images will be analyzed using automated edge detection software (Medical Imaging Applications), while intensity weighted velocity spectra segments will be saved to the GE Logiq 7 hard drive for off-line blood velocity waveform analysis. P.I. has utilized the traditional method of brachial artery flow-mediated dilation (FMD) induced by reactive hyperemia to assess vascular endothelial function in populations ranging from young healthy adults to older adults with pathological conditions.

Spygmocor - Pulse Wave Velocity (PWV) - A Spygmocor® device will be used at baseline and following each protocol to assess PWV. PWV analysis provides a non-invasive assessment of arterial stiffness. Increased arterial stiffness is known to be associated with cardiovascular disease. The participant is required to lie in a resting position for approximately 30-45 minutes. The research assistant will place ECG electrode sensors at the carotid, femoral, radial and distal artery locations. A highly sensitive pen-like device, called a tonometer, is then gently applied to record the velocity of the blood flow between each of the points.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD (GOLD stages II-IV) and matched healthy controls
* Caucasian or African American
* Both men and women
* Current and former smokers

Exclusion Criteria:

* GOLD Stage I
* Clinical diagnosis of heart disease, hypertension, or metabolic disease
* Vasoactive medications (i.e. nitrates, beta-blockers, ACE inhibitors, Viagra, etc.)
* Pulmonary hypertension
* Hypothyroidism
* Hyper-homocysteinemia
* Interstitial lung disease
* Phenylketonuria
* Pregnancy
* Sleep apnea
* Anemia
* Raynod's phenomenon
* Gangrene of the digits
* History of low platelets or coagulopathies
* Aspirin sensitivity or allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan A Harris, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Selvaraj CL, Gurm HS, Gupta R, Ellis SG, Bhatt DL. Chronic obstructive pulmonary disease as a predictor of mortality in patients undergoing percutaneous coronary intervention. Am J Cardiol. 2005 Sep 15;96(6):756-9. doi: 10.1016/j.amjcard.2005.05.016. PMID 16169353
- [Background] Anthonisen NR, Connett JE, Enright PL, Manfreda J; Lung Health Study Research Group. Hospitalizations and mortality in the Lung Health Study. Am J Respir Crit Care Med. 2002 Aug 1;166(3):333-9. doi: 10.1164/rccm.2110093. PMID 12153966
- [Background] Schachinger V, Britten MB, Zeiher AM. Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease. Circulation. 2000 Apr 25;101(16):1899-906. doi: 10.1161/01.cir.101.16.1899. PMID 10779454
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Wheatcroft SB, Williams IL, Shah AM, Kearney MT. Pathophysiological implications of insulin resistance on vascular endothelial function. Diabet Med. 2003 Apr;20(4):255-68. doi: 10.1046/j.1464-5491.2003.00869.x. PMID 12675638
- [Background] Knowles RG, Moncada S. Nitric oxide synthases in mammals. Biochem J. 1994 Mar 1;298 ( Pt 2)(Pt 2):249-58. doi: 10.1042/bj2980249. No abstract available. PMID 7510950
- [Background] Green D. Point: Flow-mediated dilation does reflect nitric oxide-mediated endothelial function. J Appl Physiol (1985). 2005 Sep;99(3):1233-4; discussion 1237-8. doi: 10.1152/japplphysiol.00601.2005. No abstract available. PMID 16103524
- [Background] Uehata A, Lieberman EH, Gerhard MD, Anderson TJ, Ganz P, Polak JF, Creager MA, Yeung AC. Noninvasive assessment of endothelium-dependent flow-mediated dilation of the brachial artery. Vasc Med. 1997;2(2):87-92. doi: 10.1177/1358863X9700200203. PMID 9546961
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Verma S, Buchanan MR, Anderson TJ. Endothelial function testing as a biomarker of vascular disease. Circulation. 2003 Oct 28;108(17):2054-9. doi: 10.1161/01.CIR.0000089191.72957.ED. No abstract available. PMID 14581384
- [Background] Maiorana A, O'Driscoll G, Taylor R, Green D. Exercise and the nitric oxide vasodilator system. Sports Med. 2003;33(14):1013-35. doi: 10.2165/00007256-200333140-00001. PMID 14599231
- [Background] Edwards DG, Schofield RS, Lennon SL, Pierce GL, Nichols WW, Braith RW. Effect of exercise training on endothelial function in men with coronary artery disease. Am J Cardiol. 2004 Mar 1;93(5):617-20. doi: 10.1016/j.amjcard.2003.11.032. PMID 14996592
- [Background] Guerci B, Kearney-Schwartz A, Bohme P, Zannad F, Drouin P. Endothelial dysfunction and type 2 diabetes. Part 1: physiology and methods for exploring the endothelial function. Diabetes Metab. 2001 Sep;27(4 Pt 1):425-34. PMID 11547216
- [Background] Zarubina EG, Mishina EA, Osadchuk MA. [The role of endothelial dysfunction in the pathogenesis of combined cardiopulmonary diseases]. Klin Med (Mosk). 2006;84(5):31-4. Russian. PMID 16827275
- [Background] Barr RG, Mesia-Vela S, Austin JH, Basner RC, Keller BM, Reeves AP, Shimbo D, Stevenson L. Impaired flow-mediated dilation is associated with low pulmonary function and emphysema in ex-smokers: the Emphysema and Cancer Action Project (EMCAP) Study. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1200-7. doi: 10.1164/rccm.200707-980OC. Epub 2007 Aug 29. PMID 17761614
- [Background] Moro L, Pedone C, Scarlata S, Malafarina V, Fimognari F, Antonelli-Incalzi R. Endothelial dysfunction in chronic obstructive pulmonary disease. Angiology. 2008 Jun-Jul;59(3):357-64. doi: 10.1177/0003319707306141. Epub 2008 Apr 2. PMID 18388072
- [Background] Eickhoff P, Valipour A, Kiss D, Schreder M, Cekici L, Geyer K, Kohansal R, Burghuber OC. Determinants of systemic vascular function in patients with stable chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Dec 15;178(12):1211-8. doi: 10.1164/rccm.200709-1412OC. Epub 2008 Oct 3. PMID 18836149
- [Background] Fukai T. Endothelial GTPCH in eNOS uncoupling and atherosclerosis. Arterioscler Thromb Vasc Biol. 2007 Jul;27(7):1493-5. doi: 10.1161/ATVBAHA.107.148239. No abstract available. PMID 17581829
- [Background] Channon KM. Tetrahydrobiopterin: regulator of endothelial nitric oxide synthase in vascular disease. Trends Cardiovasc Med. 2004 Nov;14(8):323-7. doi: 10.1016/j.tcm.2004.10.003. PMID 15596110
- [Background] Heitzer T, Brockhoff C, Mayer B, Warnholtz A, Mollnau H, Henne S, Meinertz T, Munzel T. Tetrahydrobiopterin improves endothelium-dependent vasodilation in chronic smokers : evidence for a dysfunctional nitric oxide synthase. Circ Res. 2000 Feb 4;86(2):E36-41. doi: 10.1161/01.res.86.2.e36. PMID 10666424
- [Background] Nandi M, Miller A, Stidwill R, Jacques TS, Lam AA, Haworth S, Heales S, Vallance P. Pulmonary hypertension in a GTP-cyclohydrolase 1-deficient mouse. Circulation. 2005 Apr 26;111(16):2086-90. doi: 10.1161/01.CIR.0000163268.32638.F4. Epub 2005 Apr 11. PMID 15824199
- [Background] Khoo JP, Zhao L, Alp NJ, Bendall JK, Nicoli T, Rockett K, Wilkins MR, Channon KM. Pivotal role for endothelial tetrahydrobiopterin in pulmonary hypertension. Circulation. 2005 Apr 26;111(16):2126-33. doi: 10.1161/01.CIR.0000162470.26840.89. Epub 2005 Apr 11. PMID 15824200
- [Background] Barnes PJ, Karin M. Nuclear factor-kappaB: a pivotal transcription factor in chronic inflammatory diseases. N Engl J Med. 1997 Apr 10;336(15):1066-71. doi: 10.1056/NEJM199704103361506. No abstract available. PMID 9091804
- [Background] De Boer WI. Cytokines and therapy in COPD: a promising combination? Chest. 2002 May;121(5 Suppl):209S-218S. doi: 10.1378/chest.121.5_suppl.209s. PMID 12010854
- [Background] Keatings VM, Collins PD, Scott DM, Barnes PJ. Differences in interleukin-8 and tumor necrosis factor-alpha in induced sputum from patients with chronic obstructive pulmonary disease or asthma. Am J Respir Crit Care Med. 1996 Feb;153(2):530-4. doi: 10.1164/ajrccm.153.2.8564092.
- [Background] Shapiro SD, Senior RM. Matrix metalloproteinases. Matrix degradation and more. Am J Respir Cell Mol Biol. 1999 Jun;20(6):1100-2. doi: 10.1165/ajrcmb.20.6.f151. No abstract available. PMID 10340927
- [Background] Read MA, Whitley MZ, Williams AJ, Collins T. NF-kappa B and I kappa B alpha: an inducible regulatory system in endothelial activation. J Exp Med. 1994 Feb 1;179(2):503-12. doi: 10.1084/jem.179.2.503. PMID 7507507
- [Background] Yin MJ, Yamamoto Y, Gaynor RB. The anti-inflammatory agents aspirin and salicylate inhibit the activity of I(kappa)B kinase-beta. Nature. 1998 Nov 5;396(6706):77-80. doi: 10.1038/23948. PMID 9817203
- [Background] Atkinson MH, Menard HA, Kalish GH. Assessment of salsalate, a nonacetylated salicylate, in the treatment of patients with arthritis. Clin Ther. 1995 Sep-Oct;17(5):827-37. doi: 10.1016/0149-2918(95)80061-1. PMID 8595635
- [Background] Bombardier C, Peloso PM, Goldsmith CH. Salsalate, a nonacetylated salicylate, is as efficacious as diclofenac in patients with rheumatoid arthritis. Salsalate-Diclofenac Study Group. J Rheumatol. 1995 Apr;22(4):617-24. PMID 7791151
- [Background] Pierce GL, Lesniewski LA, Lawson BR, Beske SD, Seals DR. Nuclear factor-kappaB activation contributes to vascular endothelial dysfunction via oxidative stress in overweight/obese middle-aged and older humans. Circulation. 2009 Mar 10;119(9):1284-92. doi: 10.1161/CIRCULATIONAHA.108.804294. Epub 2009 Feb 23. PMID 19237660
- [Background] Halliwell B. Free radicals and antioxidants: a personal view. Nutr Rev. 1994 Aug;52(8 Pt 1):253-65. doi: 10.1111/j.1753-4887.1994.tb01453.x. PMID 7970288
- [Background] Celermajer DS, Adams MR, Clarkson P, Robinson J, McCredie R, Donald A, Deanfield JE. Passive smoking and impaired endothelium-dependent arterial dilatation in healthy young adults. N Engl J Med. 1996 Jan 18;334(3):150-4. doi: 10.1056/NEJM199601183340303. PMID 8531969
- [Background] Celermajer DS, Sorensen KE, Georgakopoulos D, Bull C, Thomas O, Robinson J, Deanfield JE. Cigarette smoking is associated with dose-related and potentially reversible impairment of endothelium-dependent dilation in healthy young adults. Circulation. 1993 Nov;88(5 Pt 1):2149-55. doi: 10.1161/01.cir.88.5.2149. PMID 8222109
- [Background] Raitakari OT, Adams MR, McCredie RJ, Griffiths KA, Celermajer DS. Arterial endothelial dysfunction related to passive smoking is potentially reversible in healthy young adults. Ann Intern Med. 1999 Apr 6;130(7):578-81. doi: 10.7326/0003-4819-130-7-199904060-00017. PMID 10189327
- [Background] Macnee W. Pathogenesis of chronic obstructive pulmonary disease. Clin Chest Med. 2007 Sep;28(3):479-513, v. doi: 10.1016/j.ccm.2007.06.008. PMID 17720039
- [Background] Rubanyi GM, Vanhoutte PM. Superoxide anions and hyperoxia inactivate endothelium-derived relaxing factor. Am J Physiol. 1986 May;250(5 Pt 2):H822-7. doi: 10.1152/ajpheart.1986.250.5.H822. PMID 3010744
- [Background] Neunteufl T, Kostner K, Katzenschlager R, Zehetgruber M, Maurer G, Weidinger F. Additional benefit of vitamin E supplementation to simvastatin therapy on vasoreactivity of the brachial artery of hypercholesterolemic men. J Am Coll Cardiol. 1998 Sep;32(3):711-6. doi: 10.1016/s0735-1097(98)00295-2. PMID 9741516
- [Background] Plantinga Y, Ghiadoni L, Magagna A, Giannarelli C, Franzoni F, Taddei S, Salvetti A. Supplementation with vitamins C and E improves arterial stiffness and endothelial function in essential hypertensive patients. Am J Hypertens. 2007 Apr;20(4):392-7. doi: 10.1016/j.amjhyper.2006.09.021. PMID 17386345
- [Background] Title LM, Cummings PM, Giddens K, Genest JJ Jr, Nassar BA. Effect of folic acid and antioxidant vitamins on endothelial dysfunction in patients with coronary artery disease. J Am Coll Cardiol. 2000 Sep;36(3):758-65. doi: 10.1016/s0735-1097(00)00809-3. PMID 10987596
- [Background] Williams TJ, Howard M, Roget J, Esmore DS. Exercise capacity after combined heart-lung transplantation. Transplant Proc. 1992 Oct;24(5):2018. No abstract available. PMID 1412956
- [Background] Richardson RS, Secher NH, Tschakovsky ME, Proctor DN, Wray DW. Metabolic and vascular limb differences affected by exercise, gender, age, and disease. Med Sci Sports Exerc. 2006 Oct;38(10):1792-6. doi: 10.1249/01.mss.0000229568.17284.ab. PMID 17019301
- [Background] Eskurza I, Myerburgh LA, Kahn ZD, Seals DR. Tetrahydrobiopterin augments endothelium-dependent dilatation in sedentary but not in habitually exercising older adults. J Physiol. 2005 Nov 1;568(Pt 3):1057-65. doi: 10.1113/jphysiol.2005.092734. Epub 2005 Sep 1. PMID 16141271
- [Background] Ueda S, Matsuoka H, Miyazaki H, Usui M, Okuda S, Imaizumi T. Tetrahydrobiopterin restores endothelial function in long-term smokers. J Am Coll Cardiol. 2000 Jan;35(1):71-5. doi: 10.1016/s0735-1097(99)00523-9. PMID 10636262
- [Background] Padilla J, Harris RA, Fly AD, Rink LD, Wallace JP. A comparison between active- and reactive-hyperaemia-induced brachial artery vasodilation. Clin Sci (Lond). 2006 Mar;110(3):387-92. doi: 10.1042/CS20050328. PMID 16356163
- [Background] Plotnick GD, Corretti MC, Vogel RA. Effect of antioxidant vitamins on the transient impairment of endothelium-dependent brachial artery vasoactivity following a single high-fat meal. JAMA. 1997 Nov 26;278(20):1682-6. PMID 9388088
- [Background] Padilla J, Harris RA, Fly AD, Rink LD, Wallace JP. The effect of acute exercise on endothelial function following a high-fat meal. Eur J Appl Physiol. 2006 Oct;98(3):256-62. doi: 10.1007/s00421-006-0272-z. Epub 2006 Aug 3. PMID 16896723
- [Background] Tsai WC, Li YH, Lin CC, Chao TH, Chen JH. Effects of oxidative stress on endothelial function after a high-fat meal. Clin Sci (Lond). 2004 Mar;106(3):315-9. doi: 10.1042/CS20030227. PMID 14561213
- [Background] Mullen MJ, Kharbanda RK, Cross J, Donald AE, Taylor M, Vallance P, Deanfield JE, MacAllister RJ. Heterogenous nature of flow-mediated dilatation in human conduit arteries in vivo: relevance to endothelial dysfunction in hypercholesterolemia. Circ Res. 2001 Feb 2;88(2):145-51. doi: 10.1161/01.res.88.2.145. PMID 11157665
- [Background] Kingwell BA, Formosa M, Muhlmann M, Bradley SJ, McConell GK. Nitric oxide synthase inhibition reduces glucose uptake during exercise in individuals with type 2 diabetes more than in control subjects. Diabetes. 2002 Aug;51(8):2572-80. doi: 10.2337/diabetes.51.8.2572. PMID 12145173
- [Background] Lieberman EH, Gerhard MD, Uehata A, Selwyn AP, Ganz P, Yeung AC, Creager MA. Flow-induced vasodilation of the human brachial artery is impaired in patients <40 years of age with coronary artery disease. Am J Cardiol. 1996 Dec 1;78(11):1210-4. doi: 10.1016/s0002-9149(96)00597-8. PMID 8960576
- [Background] Harris RA, Nishiyama SK, Wray DW, Tedjasaputra V, Bailey DM, Richardson RS. The effect of oral antioxidants on brachial artery flow-mediated dilation following 5 and 10 min of ischemia. Eur J Appl Physiol. 2009 Nov;107(4):445-53. doi: 10.1007/s00421-009-1147-x. Epub 2009 Aug 11. PMID 19669786
- [Background] Bleeker MW, Kooijman M, Rongen GA, Hopman MT, Smits P. Preserved contribution of nitric oxide to baseline vascular tone in deconditioned human skeletal muscle. J Physiol. 2005 Jun 1;565(Pt 2):685-94. doi: 10.1113/jphysiol.2005.085936. Epub 2005 Mar 31. PMID 15802292
- [Background] Mercier JG, Hokanson JF, Brooks GA. Effects of cyclosporine A on skeletal muscle mitochondrial respiration and endurance time in rats. Am J Respir Crit Care Med. 1995 May;151(5):1532-6. doi: 10.1164/ajrccm.151.5.7735611.
- [Background] Casaburi R. Skeletal muscle function in COPD. Chest. 2000 May;117(5 Suppl 1):267S-71S. doi: 10.1378/chest.117.5_suppl_1.267s-a. PMID 10843945
- [Background] Harris RA, Padilla J, Rink LD, Wallace JP. Variability of flow-mediated dilation measurements with repetitive reactive hyperemia. Vasc Med. 2006 Feb;11(1):1-6. doi: 10.1191/1358863x06vm641oa. PMID 16669406
- [Background] Harris RA, Padilla J, Hanlon KP, Rink LD, Wallace JP. Reproducibility of the flow-mediated dilation response to acute exercise in overweight men. Ultrasound Med Biol. 2007 Oct;33(10):1579-85. doi: 10.1016/j.ultrasmedbio.2007.04.014. Epub 2007 Jun 27. PMID 17590500
- [Background] Vogel RA, Corretti MC, Plotnick GD. Effect of a single high-fat meal on endothelial function in healthy subjects. Am J Cardiol. 1997 Feb 1;79(3):350-4. doi: 10.1016/s0002-9149(96)00760-6. PMID 9036757
- [Background] Sander M, Chavoshan B, Victor RG. A large blood pressure-raising effect of nitric oxide synthase inhibition in humans. Hypertension. 1999 Apr;33(4):937-42. doi: 10.1161/01.hyp.33.4.937. PMID 10205227
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Bailey DM, Davies B, Young IS, Jackson MJ, Davison GW, Isaacson R, Richardson RS. EPR spectroscopic detection of free radical outflow from an isolated muscle bed in exercising humans. J Appl Physiol (1985). 2003 May;94(5):1714-8. doi: 10.1152/japplphysiol.01024.2002. Epub 2003 Mar 7. PMID 12626489
- [Derived] Rodriguez-Miguelez P, Gregg J, Seigler N, Bass L, Thomas J, Pollock JS, Sullivan JC, Dillard TA, Harris RA. Acute Tetrahydrobiopterin Improves Endothelial Function in Patients With COPD. Chest. 2018 Sep;154(3):597-606. doi: 10.1016/j.chest.2018.04.028. Epub 2018 Apr 26. PMID 29705218

RESULTS

PARTICIPANT FLOW:
Groups:
- COPD: AOC First, Then Placebo: Patients with COPD
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) were assessed at baseline and 2 hours following ingestion of an oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.
  After a minimum of 2 days washout, patients returned to perform all measures again but were given microcrystalline cellulose capsules as a placebo.
- COPD: Placebo First, Then AOC: Patients with COPD
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) was assessed at baseline and 2 hours following ingestion of microcrystalline cellulose capsules as a placebo.
  After a minimum of 2 days washout, patients returned to perform all measures again but were given an oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.
- Controls: AOC First, Then Placebo: Healthy age- and sex- matched controls
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) were assessed at baseline and 2 hours following ingestion of an oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.
  After a minimum of 2 days washout, subjects returned to perform all measures again but were given microcrystalline cellulose capsules as a placebo.
- Controls: Placebo First, Then AOC: Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) was assessed at baseline and 2 hours following ingestion of microcrystalline cellulose capsules as a placebo.
  After a minimum of 2 days washout, subjects returned to perform all measures again but were given an oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.
Period: First Intervention (1 Day)
Arm/Group | COPD: AOC First, Then Placebo | COPD: Placebo First, Then AOC | Controls: AOC First, Then Placebo | Controls: Placebo First, Then AOC
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Washout (2-7 Days)
Arm/Group | COPD: AOC First, Then Placebo | COPD: Placebo First, Then AOC | Controls: AOC First, Then Placebo | Controls: Placebo First, Then AOC
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | COPD: AOC First, Then Placebo | COPD: Placebo First, Then AOC | Controls: AOC First, Then Placebo | Controls: Placebo First, Then AOC
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All COPD Patients: Patients with COPD
- All Controls: Healthy age- and sex- matched controls
- Total: Total of all reporting groups
Arm/Group | All COPD Patients | All Controls | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 66 (2) | 66 (2) | 66 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 15 | 30
Height [Mean (Standard Deviation); unit: cm] | 169 (2) | 166 (2) | 168 (2)

OUTCOME MEASURES:

1. Primary Outcome: Flow-Mediated Dilation (FMD)
Description: Brachial artery FMD induced by reactive hyperemia will be used to assess vascular endothelial function at baseline and several hours after each experimental intervention.
Time Frame: Post FMD was taken approximately 110 min after baseline
Population: Participants included patients diagnosed with COPD and healthy age-matched controls.
Measure: Mean (Standard Deviation); unit: percentage of change in FMD
Arm/Group | All COPD Patients | All Controls
Number analyzed (Participants) | 30 | 30
percentage of change in FMD
  Placebo | 3.1 (0.5) | 6.7 (0.6)
  AOC Treatment | 4.7 (0.6) | 6.9 (0.7)
Statistical Analysis 1: Comparison: All COPD Patients; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: All Controls; Test type: Superiority or Other; p > 0.05, ANOVA

2. Secondary Outcome: Pulse Wave Velocity
Description: A measure of vascular stiffness at baseline and several hours after each experimental intervention.
Time Frame: Post PWV was taken approximately 90 min after baseline
Population: Patients diagnosed with COPD compared to healthy age-matched controls.
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- All COPD Patients: Patients with COPD
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) will be assessed at baseline and 2 hours following ingestion of a single oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid
- All Controls: Healthy age- and sex- matched controls
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) will be assessed at baseline and 2 hours following ingestion of a single oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid
Arm/Group | All COPD Patients | All Controls
Number analyzed (Participants) | 30 | 30
m/sec
  Placebo | 14 (1) | 11 (2)
  AOC Treatment | 11 (1) | 10 (1)
Statistical Analysis 1: Comparison: All COPD Patients; Test type: Superiority or Other; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: All Controls; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Groups:
- COPD Patients: Patients with COPD
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) will be assessed at baseline and 2 hours following ingestion of a single oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid
- Controls: Healthy age- and sex- matched controls
  Brachial artery flow-mediated dilation, direct assessment of oxidative stress via EPR spectroscopy (O2-) and biomarkers of oxidative stress (8-isoprostane, LH, SOD) will be assessed at baseline and 2 hours following ingestion of a single oral antioxidant cocktail (1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid.) Antioxidant Cocktail: 1g of vitamin C, 600 IU of vitamin E, and 600 mg of alpha-lipoic acid
Arm/Group | COPD Patients | Controls
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No